CLINICAL TRIAL: NCT03249324
Title: Preventing Obesity in Military Communities: Mother-Baby
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Collaborators: Naval Hospital Camp Lejeune (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NHCL.2012.0011
Record Dates: First submitted 2017-06-20; First posted 2017-08-15 (Actual); Last update posted 2017-08-15 (Actual); Status verified 2017-08

CONDITIONS: Pregnancy; Overweight; Obesity
Keywords: Pregnancy; Overweight; Obesity; Prevention; Positive-gain counseling
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Positive-Gain Counseling (PGC) (Experimental): Positive-gain-based health promotion interventions capitalize on the basic human desire to maintain consistency between one's words and actions for beneficial outcomes. Participants will discuss potential costs of unhealthy behaviors and the benefits of healthier lifestyle choices, and how they apply not only to adults, but also to developing children. Theoretically, discussing these perspectives will make the mothers more likely to make healthier lifestyle choices in the future.
  Interventions: Behavioral: Positive-Gain Counseling (PGC)
- Usual Care (UC) (Active Comparator): UC includes regular clinic visits, routine blood and urine screening tests, and anticipatory guidance from a primary care provider in accordance with the VA/DoD Guideline for the Management of Pregnancy. After delivery, participants receive routine well-child care in accordance with established guidelines from the American Academy of Pediatrics and the American Academy of Family Physicians.
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Positive-Gain Counseling (PGC) — Positive-gain-based health promotion interventions capitalize on the basic human desire to maintain consistency between one's words and actions for beneficial outcomes. Participants will be asked to discuss potential adverse effects of obesity, an unhealthy diet, and sedentary behavior, as well as the benefits of maintaining a physically fit body, eating a healthy diet, and regular physical activity. They will also discuss the costs and benefits as they apply to developing children. Theoretically, discussing and reviewing these perspectives will make the mothers more apt to make healthier lifestyle choices in the future. Women randomized to the positive-gains counseling (PGC) group will have PGC sessions once during each trimester and at 2 weeks, 2 months, 4 months and 6 months postpartum. PGC participants will also receive prenatal care in accordance with the VA/DoD Guideline for the Management of Pregnancy.
  Arms: Positive-Gain Counseling (PGC)
Other: Usual Care — Women in the usual care (UC) group will receive prenatal care in accordance with the VA/DoD Guideline for the Management of Pregnancy. This entails regular clinic visits, routine blood and urine screening tests, and anticipatory guidance. Routine well-child care appointments will take place at 2-3 days, 2 weeks, 2 months, 4 months, 6 months, 9 months and 12 months after birth. During routine well-child visits, height, weight, and vital signs are measured, developmental milestones are reviewed, and a thorough physical examination is performed. Age-appropriate immunizations are provided as is parental anticipatory guidance, including the importance of breastfeeding. Participants enrolled in the UC group will receive anticipatory guidance from their primary care provider in the usual fashion. Providers will deliver this anticipatory guidance with no external cues or counseling provided by the research team.
  Arms: Usual Care (UC)

SUMMARY:
Women with pre-pregnancy obesity, women who exceed recommended weight gain during pregnancy, and children who experience rapid and excess growth during the first year of life are all at risk for subsequent obesity. The purpose of this study is to examine creative cognitive strategies to promote healthy weight gain during pregnancy, creating a sound substrate of metabolic programming for the critical first six months of life. A trans-disciplinary approach utilizing a patient- and family-centered intervention and active patient engagement with counseling for positive gain will work with women to shape lifestyle during pregnancy and postpartum, and when feeding their infants in the first 6 months of life. It is hypothesized patient engagement with counseling for positive gains will successfully mitigate excess weight gain in both pregnancy and infancy compared to usual care. Moreover, data will be examined to assess whether psychological variables, work and school climate, and social support factors influence body weight gain trajectories and/or weight loss during and after pregnancy.

DETAILED DESCRIPTION:
Obesity is increasingly common among reproductive aged women and women presenting for their first pregnancy. Women with overweight and obesity are more likely to exceed recommended weight gain during pregnancy and retain excess weight after delivery. Women with pre-pregnancy obesity, women who exceed recommended weight gain during pregnancy, and children who experience rapid and excess growth during the first year of life are all at risk for subsequent obesity. Additionally, maternal obesity is a significant risk factor for pregnancy complications (i.e., hypertensive disorders of pregnancy, gestational diabetes) and is associated with adverse pregnancy outcomes, including excess fetal weight at birth. The goal of this study is to test the effectiveness of active patient engagement with counseling for positive gain to mitigate excess weight gain in women during pregnancy and postpartum, and in the first six months of life. Pregnant women eligible to receive care in the Military Health System (MHS) will be randomized to receive either the positive-gain counseling (PGC) prevention program or usual care (UC). PGC is designed to empower women to examine food choices and activity patterns during pregnancy to help them adhere to the Institute of Medicine (IOM) recommended weight gain standards. PGC patients will be paired with counselors who follow their pregnancy from start to finish, as well as providing neonatal and infant support in a continuous fashion as part of team-based care. Women in the usual care (UC) group will receive prenatal care in accordance with the VA/DoD Guideline for the Management of Pregnancy. Both groups will receive routine well-child care in accordance with established guidelines from the American Academy of Pediatrics and the American Academy of Family Physicians. Routine well-child care appointments (UC) take place at 2-3 days after birth, 2 weeks of life, 2 months of life, 4 months, 6 months, 9 months and 12 months. Participants' weight status, food intake, and mood will be assessed once during each trimester and at 2 weeks, 2 months, 4 months, and 6 months postpartum. Individuals enrolled in the PGC group will receive specific counseling once during each trimester and at 2 weeks, 2 months, 4 months and 6 months postpartum. Well-child sessions will focus on positive-gain-based cognitive strategies to promote breastfeeding, recognition of satiety cues and other healthy food choices. It is hypothesized that participants who receive the positive-gains counseling program will show significantly less weight gain in both pregnancy and infancy relative to those randomized to usual care.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 35 years
* Absence of underlying medical conditions that would place the pregnancy in the high-risk category (e.g., hypertension, pre-existing diabetes mellitus, thyroid disease, multiple gestations)
* Baseline BMI (on determination of pregnancy) >18 kg/m2 and ≤29.9 kg/m2
* Plan to reside in the study area (Jacksonville, NC area) for at least 18 months
* Eligible for care within the Military Health System (MHS)
* No planned surgeries, medical interventions, or other procedures that would place participants in the high-risk pregnancy category
* No involvement in a commercial or military weight management program in the past 3 months
* Fluent command of the English language

Exclusion Criteria:

* Current involvement in a structured weight loss program
* BMI of ≤18 kg/m2 or ≥30 kg/m2
* Potential participants with high-risk pregnancies. Participants will be placed in the high risk pregnancy category if they have any underlying medical conditions (e.g. hypertension, diabetes, thyroid disease, multiple gestations) placing the subject into a high-risk category by American College of Obstetrics and Gynecology (ACOG) standards
* Planned surgeries or other procedures that would place participants in the high-risk pregnancy category

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2014-11; Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Maternal weight gain | Pre-pregnancy to delivery

SECONDARY OUTCOMES:
Infant birth weight | Birth
  Data will be collected from the participant's inpatient medical records (Essentris) at Naval Hospital Camp Lejeune
Development of gestational diabetes | Gestation
  Data will be collected for all participants from the outpatient electronic medical records (AHLTA) at Naval Hospital Camp Lejeune
Need for induction of labor and methods of labor induction used | Labor and delivery
  Data will be collected from the participant's inpatient medical records (Essentris) at Naval Hospital Camp Lejeune
Mode of Delivery | Birth
  Mode of delivery (e.g., vaginal or Caesarean section) will be collected from the participant's inpatient medical records (Essentris) at Naval Hospital Camp Lejeune
Length of Labor | Onset of latent phase of labor to delivery of the placenta and fetal membranes
  The length of labor will be collected from the participant's inpatient medical records (Essentris) at Naval Hospital Camp Lejeune
Need for anesthesia or analgesics and forms of anesthesia or analgesics used during labor | Labor and delivery
  Data will be collected from the participant's inpatient medical records (Essentris) at Naval Hospital Camp Lejeune

CONTACTS AND LOCATIONS:
Overall Officials: Mark Stephens, MD, Principal Investigator — Uniformed Services University of the Health Sciences; Linda Chan, MD, Principal Investigator — Naval Hospital Camp Lejeune
Locations (1):
- Naval Hospital Camp Lejeune, Marine Corps Base Camp Lejeune, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No